CLINICAL TRIAL: NCT04052373
Title: Surgical Peri-implantitis Treatment With and Without Implantoplasty
Brief Title: Peri-implantitis Implantoplasty Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Anders Verket, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMPLANTOPLASTY
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peri-implantitis treatment with implantoplasty (Experimental): Open flap debridement with implantoplasty treatment
  Interventions: Procedure: Implantoplasty; Procedure: Open flap debridement alone
- Peri-implantitis treatment without implantoplasty (Active Comparator): Open flap debridement withput implantoplasty treatment
  Interventions: Procedure: Implantoplasty; Procedure: Open flap debridement alone

INTERVENTIONS:
Procedure: Implantoplasty — Implantoplasty is the mechanical smoothening of rough titanium implants as part of the surgical treatment of peri-implantitis. Treatment is thought to facilitate self-performed oral hygiene.
Procedure: Open flap debridement alone — Open flap debridement alone

SUMMARY:
This double arm, split-mouth, single centre, controlled, randomised clinical study is designed to examine the effect of implantoplasty in treatment of peri-implantitis.

Peri-implantitis will be treated with open flap debridement, with or without implantoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Peri-implantitis (according to 2018 criteria) on minimum 2 implants of similar surface and defect type
* Competent to give consent
* Exposed, modified implant surface with loss >2mm

Exclusion Criteria:

* Previous radiotherapy to the jaws, current use of chemotherapy, systemic long-term corticosteroid treatment
* Present or past use of bisphosphonate treatment • Pregnant or nursing subjects
* Patients classified as > class II according to ASA classification
* Implant unavailable for implantoplasty treatment
* Inhability to comprehend and respond to the quality of life questionnaire
* Examiners/operators deem original placement of implant (angle, position) suboptimal and considered to play a major role in development of peri-implantitis
* History of peri-implantitis surgery prior to 6 months of screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing | 12 months after treatment
  Measured with a periodontal probe
Bleeding on probing | 24 months after treatment
  Measured with a periodontal probe

SECONDARY OUTCOMES:
Suppuration | 12 months after treatment
  Visible suppuration upon probing the implant with a periodontal probe
Suppuration | 24 months after treatment
  Visible suppuration upon probing the implant with a periodontal probe
Pocket probing depth | 12 months after treatment
  Measured with a periodontal probe
Pocket probing depth | 24 months after treatment
  Measured with a periodontal probe
Changes in patient-reported quality of life (QoL) | Preoperatively compared to 24 months after treatment
  To assess QoL changes related to mouth and teeth prior to therapy to after therapy by the use of "The Oral Impacts on Daily Performance (OIDP)" instrument. Each question is assessed by a 5-point scale; (1) never affected; (2) less than once a month; (3) once or twice a month; (4) once or twice a week; and (5) every or nearly every day. The higher number represents more severe impact on quality of life; e.g. worse outcome.
  Each item will be dichotomised yielding the categories (A) affected; including scale categories (2)-(5), and (B) unaffected; including category (1)
Clinical attachment loss measurements | 12 months after treatment
  Measured with a periodontal probe
Clinical attachment loss measurements | 24 months after treatment
  Measured with a periodontal probe
Radiographic bone loss | 12 months after treatment
  Measured on standardized radiograps
Radiographic bone loss | 24 months after treatment
  Measured on standardized radiograps
Implant fracture | 24 months
  Clinical examination to assess whether implants have fractured following treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Institute of Clinical Dentistry, Faculty of Dentistry, University of Oslo, Oslo
  - Institute of Clinical Dentistry, University of Oslo, Norway, Oslo